CLINICAL TRIAL: NCT04230083
Title: Bioavailability of a Formulation of Dienogest 2.0 mg Coated Tablets With Regards to the Marketed Reference Product
Brief Title: Bioavailability of Dienogest 2.0 mg With Regards to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP8820-01
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Bioequivalence
MeSH Terms: interventions — dienogest; Drug Evaluation; Patents as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dienogest Test Product (Experimental): Participants will receive one tablet of the test formulation containing Dienogest 2.0 mg. The tablets will be taken with water.
  Interventions: Drug: Dienogest 2.0 mg Test Drug
- Dienogest Reference Product (Active Comparator): Participants will receive one tablet of the test formulation containing Dienogest 2.0 mg. The tablets will be taken with water.
  Interventions: Drug: Dienogest 2.0 mg Reference Product

INTERVENTIONS:
Drug: Dienogest 2.0 mg Test Drug — Bioequivalence
  Other Names: Investigational Medicinal Product
  Arms: Dienogest Test Product
Drug: Dienogest 2.0 mg Reference Product — Bioequivalence
  Other Names: Visannette (Trademark)
  Arms: Dienogest Reference Product

SUMMARY:
This Pivotal study will investigate the bioavailability in women of 1 tablet formulations containing Dienogest 2.0 mg. The Pivotal study will be performed at a single site with 30 subjects. Participants will take 1 tablet of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There will be a washout of at least 14 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of Dienogest of 1 tablet formulation with Dienogest 2.0 mg and to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Laboratorios Andrómaco S.A.
* Reference Product: Visannette [Trademark], product of Bayer AG, Germany. The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters area under the plasma concentration-time curve from time zero to time t (AUC0-t) and from time zero to 72 hours (AUC0-72), and maximum plasma concentration (Cmax) for total Dienogest will be determined. Participants will be confined in the study site for approximately 36 hours during each study period (for 12 hours pre-dosing and for 24 hours post dosing) during which pharmacokinetic (PK) blood samples will be obtained. 16 blood samples will be taken up to 24 hours after the administration in each period. Participants will return to the site to provide additional blood samples at 48 h, and 72 h postdose.

The washout period between the two study periods will be at least 14 days. The samples from each participant will be analyzed with 2 methods of highperformance liquid chromatography-tandem mass spectrometry bioanalytical assays to quantify total Dienogest in plasma.

The safety objective is to evaluate the tolerability of both formulations in women by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant and non-breastfeeding women
* Women of childbearing age with an acceptable form of contraception during the study
* 18 to 55 years old inclusive; BMI greater than or equal to 18.51 and less than or equal to 29.99
* Non-smoking or smoke only 3 cigarettes every 7 days
* With results of laboratory tests, electrocardiogram and chest radiography in normal and / or negative or abnormal ranges but without clinical relevance and declared suitable for study by the doctor after the physical examination
* Capable to understand the Informed Consent Form

Exclusion Criteria:

* Study site or sponsor staff or family members
* With history of drug and/or alcohol abuse
* Smokers more tan 3 cigarettes every 7 days
* Vitamin supplements intake 7 days prior to the administration of the medications under study
* Any recent change in eating habits or physical exercise
* Using of a pharmacological therapy (except over the counter medication use 7 days prior to the study)
* Hypersensitivity to the study drug or to other chemically related compounds, history of serious adverse reactions or hypersensitivity to any medication
* Use, during the 28 days prior to the start of the study, of medications known to alter liver enzyme activity
* Consumption of beverages or food containing grapefruit or pink grapefruit, within 7 days prior to each administration of the study medication and consumption of alcohol, caffeine or beverages or foods containing xanthines 24 hours before each administration of the study medication until the last sample of each period
* History of any significant cardiovascular disease
* Acute disease that generates significant physiological changes from the time of selection until the end of the study
* HIV, Hepatitis B and/or C positive
* Presence or history of thrombophlebitis, thrombosis or thromboembolic disorders, deep vein thrombosis, pulmonary embolism or known coagulopathy.
* Donation or loss of a significant volume (more than 100 mL) of blood or plasma or platelets during the 3 months prior to the start of the study
* Subjects who have participated in any type of clinical study during the 3 months prior to the start of the study
* History of any gastrointestinal surgery that could affect drug absorption
* Presence of fainting history or fear to blood collection

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Total Dienogest: area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) | From tablet intake and up to 72 hours after tablet intake
  20 samples up to 72 hours will be taken after the administration in each period.
Total Dienogest: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | From tablet intake and up to 72 hours after tablet intake
  20 samples up to 72 hours will be taken after the administration in each period.
Total Dienogest: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  20 samples up to 72 hours will be taken after the administration in each period.
Total Dienogest: Time to achieve maximum plasma concentration (tmax) | From tablet intake and up to 72 hours after tablet intake
  20 samples up to 72 hours will be taken after the administration in each period.

CONTACTS AND LOCATIONS:
Locations (1):
- Innolab, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No